CLINICAL TRIAL: NCT02266589
Title: Research of Little Doses of Hydrocortisone on Coagulation Dysfunction in Patients With Septic Shock
Brief Title: Stress Doses of Hydrocortisone on Coagulation Dysfunction in Patients With Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Nanjing PLA General Hospital, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011NLY031
Record Dates: First submitted 2014-10-12; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Septic Shock; Sepsis
Keywords: coagulopathy; hydrocortisone; organ failure; hemodynamic improvement induced by hydrocortisone
MeSH Terms: conditions — Shock, Septic; Sepsis; Hemostatic Disorders | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone (Experimental): little doses of hydrocortisone
  Interventions: Drug: Hydrocortisone
- Placebo (No Intervention): Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone hemisuccinate (Roussel-Uclaf, Romainville, France), 50 mg intravenously every 6 hrs
  Arms: Hydrocortisone

SUMMARY:
The purpose of this study is to find out whether stress doses of hydrocortisone attenuate coagulation dysfunction in patients with septic shock. And discuss the probable mechanism by which little doses of hydrocortisone influence coagulation system in sepsis.

DETAILED DESCRIPTION:
Patients were randomized to receive either low-dose hydrocortisone or matching placebo.Severity of coagulopathy was estimated using ISTH DIC score. We determined the complications and mortality in two groups, and analyzed the relationship between hydrocortisone and coagulopathy.

ELIGIBILITY:
Inclusion Criteria:

* All patients(age≧18y)
* Admitted for septic shock were considered eligible if they had no life-threatening systemic disease (ASA groups 1~3)

Exclusion Criteria:

* Lactation
* Mental disorders
* Disseminated cancer
* Secondary cancers
* Inflammatory bowel disease, or diseases hindering epidural analgesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
coagulopathy | 30 days after inclusion
  ISTH score

SECONDARY OUTCOMES:
death | 30 days after inclusion
clinical complications | 30 days after inclusion
  MODS SOFA score